CLINICAL TRIAL: NCT01480388
Title: A Phase 2b Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel-group, Dose Range Finding Study of JNJ-39758979 in Subjects With Active Rheumatoid Arthritis Despite Concomitant Methotrexate Therapy
Brief Title: A Dose Range Finding Study of JNJ-39758979 in Patients With Active Rheumatoid Arthritis Currently Treated With Methotrexate
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated prematurely due to 2 cases of agranulocytosis in a different clinical trial with this same drug.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR018814; 39758979ARA2001 (Other: Janssen Research & Development, LLC); 2011-002849-36 (EudraCT Number)
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Active Rheumatoid Arthritis; Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Swollen and tender joints; Dose range finding study; Concurrent treatment with methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo/JNJ-39758979 (300 mg/d)
- JNJ-39758979 (10 mg/d) (Experimental)
  Interventions: Drug: JNJ-39758979 (10 mg)
- JNJ-39758979 (30 mg/d) (Experimental)
  Interventions: Drug: JNJ-39758979 (30 mg)
- JNJ-39758979 (100 mg/d) (Experimental)
  Interventions: Drug: JNJ-39758979 (100 mg)
- JNJ-39758979 (300 mg/d) (Experimental)
  Interventions: Drug: JNJ-39758979 (300 mg)

INTERVENTIONS:
Drug: Placebo/JNJ-39758979 (300 mg/d) — Form = tablet, route = oral adminstration placebo once daily from Week 0 to Week 24 followed by JNJ-39758979 300 mg once daily from Week 24 to Week 48.
  Other Names: Inactive medical substance
  Arms: Placebo
Drug: JNJ-39758979 (10 mg) — Form = tablet, route = oral adminstration once daily up to 48 weeks
  Arms: JNJ-39758979 (10 mg/d)
Drug: JNJ-39758979 (30 mg) — Form = tablet, route = oral adminstration once daily up to 48 weeks
  Arms: JNJ-39758979 (30 mg/d)
Drug: JNJ-39758979 (100 mg) — Form = tablet, route = oral adminstration once daily up to 48 weeks
  Arms: JNJ-39758979 (100 mg/d)
Drug: JNJ-39758979 (300 mg) — Form = tablet, route = oral adminstration once daily for 48 weeks
  Arms: JNJ-39758979 (300 mg/d)

SUMMARY:
The purpose of the study is to assess the efficacy, safety and tolerability of JNJ-39758979 at doses of 10, 30, 100, and 300 mg/day compared with placebo (inactive medical substance) in patients with active rheumatoid arthritis despite concomitant treatment with methotrexate (MTX).

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor patient knows if the patient is receiving JNJ-39758979 or placebo), multicenter, randomized (patients are assigned to treatment by chance), placebo-controlled, dose range finding study of JNJ-39758979 in patients with stable methotrexate treatment through Week 24. The study will consist of 4 periods: a screening period, a 24-week placebo-controlled period, a 24-week extension period, and a 5-week safety follow-up period. The duration of participation in the study for an individual patient will be up to 59 weeks (including screening). All patients will be randomly assigned in a 1:1:1:1:1 ratio to receive placebo or JNJ-39758979 10 mg, 30 mg, 100 mg, or 300 mg once daily. At Week 24, all patients remaining in the placebo group will start to receive JNJ-39758979 300 mg/day. Safety assessments and evaluations to determine the efficacy of JNJ-39758979 to reduce the signs and symptoms of rheumatoid arthritis will be performed at study visits. The extension and safety follow-up periods of this study will continue through Week 53 in order to assess the safety and for maintenance of efficacy of patients.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of rheumatoid arthritis (RA) for at least 6 months before screening.
* Positive test for either anti-cyclic citrullinated peptide (anti-CCP) antibody or rheumatoid factor (RF) in serum at screening.
* Has active RA defined as persistent disease activity with the following criteria: at least 6 swollen and 6 tender joints, and serum CRP ≥ 0.70 mg/dL at screening.
* Has been treated with and tolerated methotrexate (MTX) treatment at dosages of 10 to 25 mg/week for a minimum of 6 months prior to screening and must be on a stable dose for a minimum of 8 weeks prior to screening
* Must be post-menopausal or if pre-menopausal, must use an acceptable form of birth control
* Has completed at least 5 days of daily pain diary in the 10 days prior to randomization.

Exclusion Criteria:

* Has inflammatory diseases other than RA, such as Lupus.
* Is currently receiving treatment for RA other than methotrexate, NSAIDS, or oral corticosteroids such as prednisone, or pain medicines.
* Has ever received any biologic agent for a rheumatic indication.
* Has current signs or symptoms of liver insufficiency or cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, psychiatric, or metabolic disturbances that are severe, progressive, or uncontrolled.
* Has moderate or severe renal insufficiency
* Has a recent (within 2 months) serious infection
* Has had an opportunistic infection.
* Has had cancer within the past 5 years (except certain skin or cervical conditions)
* Has abused substances or alcohol within the past 2 years
* Has active Hepatitis B or C infection
* Has had active tuberculosis
* Has had exposure to tuberculosis without preventative treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The primary end point is change from baseline in Disease Activity Score 28 (DAS28) (CRP) at Week 12 | Baseline, Week 12

SECONDARY OUTCOMES:
Change from baseline in DAS28 (CRP) at Week 24 | Baseline, Week 24
Change from baseline in DAS28 (ESR) at Week 12 and Week 24 | Baseline, Week 12 and Week 24
DAS28 (CRP) response rates at Week 12 and Week 24 | Week 12, Week 24
DAS28 (ESR) response rates at Week 12 and Week 24 | Week 12, Week 24
DAS28 (CRP) remission rates at Week 12 and Week 24 | Week 12, Week 24
American college of rheumatology (ACR) 20/50/70 response rates at Week 12 and Week 24 | Week 12, Week 24
Hybrid ACR response at Week 12 and Week 24 | Week 12, Week 24
ACR/European League Against Rheumatism (EULAR) remission rates at Week 12 and Week 24 | Week 12, Week 24
Change from baseline in Simplified Disease Activity Index (SDAI) at Week 12 and Week 24 | Baseline, Week 12, Week 24
Change from baseline in Clinical Disease Activity Index (CDAI) at Week 12 and Week 24 | Baseline, Week 12, Week 24
Health Assessment Questionnaire - Disability Index (HAQ-DI) response at Week 12 and Week 24 | Week 12, Week 24
Change from baseline in HAQ-DI score at Week 12 and Week 24 | Baseline, Week 12 and Week 24
Percent change from baseline in ESR levels at Week 12 and Week 24 | Baseline, Week 12 and Week 24
Percent change from baseline in ACR components at Week 12 and Week 24 | Baseline, Week 12 and Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Development, L.L.C. Clinical Trial, Study Director — Janssen Research & Development, LLC